CLINICAL TRIAL: NCT01800786
Title: Memory Consolidation in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ina E. Donlagic, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OSAM; K23HL103850-01 (NIH)
Record Dates: First submitted 2013-02-23; First posted 2013-02-28 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSA-CPAP group (Active Comparator): OSA patient will use CPAP for 3 months
  Interventions: Device: CPAP
- OSA -no CPAP (No Intervention): newly diagnosed OSA patient will not wear CPAP for 3 months

INTERVENTIONS:
Device: CPAP
  Arms: OSA-CPAP group

SUMMARY:
The overarching goal of the research proposed here is to test the hypothesis (i) that the pathophysiological mechanisms of OSA lead to deterioration in sleep-dependent memory consolidation across memory systems, with the genetic marker APOε4 as a modulator, and (ii) that CPAP can reverse some or all of these measured memory deficits.

In addition, we are exploring which aspects of OSA (e.g., changes in sleep architecture, measures of hypoxemia, or the EEG power spectrum) most likely impact sleep-dependent memory processing.To this end, we are using specific cognitive tasks for which sleep-dependent memory consolidation processes have previously been demonstrated by our group and others. In addition, we are carrying out quantitative EEG power spectral analyses, to delineate abnormal functioning of brain regions with more precision.

ELIGIBILITY:
Subject selection

General inclusion criteria:

* Men and women ages 18 to 80 years old
* Good health as determined by a medical and psychiatric history and physical examination
* An absence of any medical or psychiatric disorders (other than OSA and treated hypertension) that could influence excessive daytime sleepiness
* The ability to complete self-rating scales and computer-based testing
* Beck Depression Inventory score ≤16
* Healthy controls will be excluded with and Epworth Sleepiness Scale (ESS) score > 10/24, OSA patients will be excluded from randomization with an ESS score >18/24.
* Subjects must agree to abstain from alcohol consumption from the day before and throughout Session 1 and Session 2.

Criteria for OSA patients:

* Newly diagnosed with OSA and with no prior exposure to CPAP
* Quantified apnea-hypopnea index greater than 5/hr (AHI, defined as the number of apneas and/or hypopneas per hour of sleep)
* Subjects must agree to limit alcohol use between Session 1 and Session 2 to one or fewer alcoholic drinks daily or up to 4 drinks weekly

Criteria for Healthy control group:

• Subjects will be matched to the obstructive sleep apnea patient group for age, race, body mass index, education and intelligence (WAIS - full scale)

Subgroup selection:

An additional subgroup of OSA patients and controls, who are taking antidepressants, will be recruited. Except for the current treatment with antidepressants all other exclusion and exclusion criteria will be applied.

The following classes of antidepressants will be eligible:

* Selective serotonin reuptake inhibitors
* Serotonin-norepinephrine reuptake inhibitors
* Noradrenergic and specific serotonergic antidepressants
* Norepinephrine-dopamine reuptake inhibitors

Exclusion criteria

ALL PARTICIPANTS:

Potential participants (OSA patients and controls) are excluded if one or more of the following conditions are found:

* Any history of clinically significant, uncontrolled medical or psychiatric condition (treated or untreated), other than OSA and hypertension (self-report)
* History of serious heart disease or renal failure (self-report)
* History of head injury (self-report)
* Inability to type (e.g., physical disability, arthritis) or to exercise
* A lifetime history of alcohol, narcotic or any other drug abuse (self-report)
* Use of medications, over-the counter drugs or nutritional supplements known to have an effect on sleep, cognition and/or daytime vigilance (self-report)
* Female subjects who are pregnant cannot take part in the study. If a female subject becomes pregnant during the study, she will have to stop participation
* Presence of any of the following sleep disorders:

  * Cheyne-Stokes breathing or central sleep apnea (> 10% of events central) (screening sleep study)
  * Circadian rhythm disorder (structured interview)
  * REM sleep without atonia or REM behavior disorder (structured interview and screening sleep study )
  * Parasomnias (structured interview)
  * PLMS index of >15/h (screening sleep study)
  * Insomnia (structured interview and 2 weeks sleep diaries)
  * Narcolepsy (structured interview)
* Left-handedness (only MSLT participants)- (self-report)
* uncorrected vision impairment and/or visual field defect (self report, screening examination)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ina Djonlagic, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- OSA-CPAP Group: OSA patient will use CPAP for 3 months
  CPAP= continuous positive airway pressure therapy
  OSA= obstructive sleep apnea
Period: Overall Study
Arm/Group | OSA-CPAP Group | OSA -no CPAP
Started | 17 | 16
Completed | 15 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OSA-CPAP Group | OSA -no CPAP | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.4) | 46.4 (13) | 47.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overnight Change in Declarative Memory Performance
Description: At 3 months, we compared average overnight changes between evening and morning performance on a declarative memory test between untreated OSA subjects and those who received CPAP therapy for 3 months.
  Positive numbers represent an increase in performance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent change in performance
Arm/Group | OSA-CPAP Group | OSA -no CPAP
Number analyzed (Participants) | 17 | 16
percent change in performance | 11.2 (0.8) | 6.5 (0.11)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | OSA-CPAP Group | OSA -no CPAP
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes